CLINICAL TRIAL: NCT03200860
Title: Randomized, Double Blind, Placebo Controlled, Multicenter Pilot Study on the Effects of Empagliflozin on Clinical Outcomes in Patients With Acute Decompensated Heart Failure (EMPA-RESPONSE-AHF)
Brief Title: Effects of Empagliflozin on Clinical Outcomes in Patients With Acute Decompensated Heart Failure
Acronym: EMPA-RESPONSE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2017-001679-22
Record Dates: First submitted 2017-06-23; First posted 2017-06-27 (Actual); Results first posted 2020-02-19 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Heart Failure Acute; Heart Failure，Congestive; Heart Failure; With Decompensation
Keywords: heart failure; diuretic response; empagliflozin
MeSH Terms: conditions — Heart Failure | interventions — empagliflozin

STUDY DESIGN:
Intervention Model Description: randomized, placebo-controlled, double-blind, parallel group, multicenter study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double blind, placebo controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Empagliflozin (Active Comparator): Empagliflozin 10 mg daily, oral, 30 days
  Interventions: Drug: Empagliflozin 10 MG
- Placebo (Placebo Comparator): Matching Placebo 10 mg daily, oral, 30 days
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Empagliflozin 10 MG — 10 mg daily, oral, 30 days
  Arms: Empagliflozin
Drug: Placebo Oral Tablet — Matching Placebo, 10 mg daily, oral, 30 days
  Arms: Placebo

SUMMARY:
Acute decompensated heart failure is the fastest growing disease in the world and the leading cause of hospital admissions worldwide. Short term mortality and rehospitalization are extremely high (20-30% within 3-6 months) and there is no therapy available that improves clinical outcome in these patients. Empagliflozin is a selective inhibitor of sodium glucose co-transporter with diuretic and renal- protective properties. In patients with type 2 diabetes at high risk for cardiovascular events, empagliflozin reduced the risk of hospitalization for heart failure by 35%. Based on the promising pharmacological profile of empagliflozin in relation to the needs for treatment of acute decompensated heart failure, we hypothesize that empagliflozin exerts positive effects in acute decompensated heart failure, with or without diabetes,

This is a randomized, placebo-controlled, double-blind, parallel group, multicenter study in subjects admitted for acute decompensated heart failure. Eighty eligible subjects will be randomized in a 1:1 ratio to receive either empagliflozin 10 mg/day or matched placebo.

DETAILED DESCRIPTION:
This is a randomized, placebo-controlled, double-blind, parallel group, multicenter study in subjects admitted for acute decompensated heart failure. Eighty eligible subjects will be randomized in a 1:1 ratio to receive either empagliflozin 10 mg/day or matched placebo.

Treatment will be continued until 30 days after index event, and primary efficacy measurements will be carried out during hospitalization and safety events until 60 days after index hospitalisation.

ELIGIBILITY:
Inclusion Criteria:

* Male or female >18 years of age; Women of non-child-bearing potential must have a documentation of surgical sterilization (hysterectomy and/or bilateral oophorectomy) OR must have experienced menopause (no menses for >12 months). Women of child bearing potential must have a negative pregnancy test, AND must use highly effective methods of contraception during treatment with IP plus 5 days after the end of study drug administration.
* Hospitalized for AHF; AHF is defined as including all of the followings measured at any time between presentation (including the emergency department) and the end of screening:

  1. Dyspnea at rest or with minimal exertion
  2. Signs of congestion, such as edema, rales, and/or congestion on chest radiograph
  3. BNP ≥350 pg/mL or NT-proBNP ≥1,400 pg/mL (for patients with AF: BNP≥500 pg/mL or NT-proBNP ≥2,000 pg/mL)
  4. Treated with loop diuretics at screening
* Able to be randomized within 24 hours from presentation to the hospital
* Able and willing to provide freely given written informed consent
* eGFR (CKD-EPI) ≥30 ml/min/1.73m2 between presentation and randomization

Exclusion Criteria:

* Diabetes Mellitus Type I
* Dyspnea primarily due to non-cardiac causes
* Cardiogenic shock
* Acute coronary syndrome within 30 days prior to randomization
* Planned or recent percutaneous or surgical coronary intervention within 30 days prior to randomization
* Signs of keto-acidosis and/or hyperosmolar hyperglaecemic syndrome (pH>7.30 and glucose >15 mmol/L and HCO3>18 mmol/L)
* Pregnant or nursing (lactating) women
* Current participation in any interventional study
* Inability to follow instructions or comply with follow-up procedures
* Any other medical conditions that may put the patient at risk or influence study results in the investigator's opinion, or that the investigator deems unsuitable for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2017-12-18 (Actual); Primary Completion 2019-09-18 (Actual); Study Completion 2019-09-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adriaan Voors, Prof. Dr., Principal Investigator — University Medical Center Groningen
Locations (5):
- Netherlands (5):
  - TREANT Zorggroep, Emmen, Drenthe
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch, North Brabant
  - ISALA Klinieken, Zwolle, Overijssel
  - Antonius Ziekenhuis, Sneek, Provincie Friesland
  - University Medical Center Groningen, Groningen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zinman B, Wanner C, Lachin JM, Fitchett D, Bluhmki E, Hantel S, Mattheus M, Devins T, Johansen OE, Woerle HJ, Broedl UC, Inzucchi SE; EMPA-REG OUTCOME Investigators. Empagliflozin, Cardiovascular Outcomes, and Mortality in Type 2 Diabetes. N Engl J Med. 2015 Nov 26;373(22):2117-28. doi: 10.1056/NEJMoa1504720. Epub 2015 Sep 17. PMID 26378978
- [Background] Wanner C, Inzucchi SE, Lachin JM, Fitchett D, von Eynatten M, Mattheus M, Johansen OE, Woerle HJ, Broedl UC, Zinman B; EMPA-REG OUTCOME Investigators. Empagliflozin and Progression of Kidney Disease in Type 2 Diabetes. N Engl J Med. 2016 Jul 28;375(4):323-34. doi: 10.1056/NEJMoa1515920. Epub 2016 Jun 14. PMID 27299675

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Empagliflozin | Placebo
Started | 41 | 39
Completed | 40 | 39
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Empagliflozin | Placebo | Total
Number analyzed (Participants) | 40 | 39 | 79
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 12 | 16
  >=65 years | 36 | 27 | 63
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 79 [73 to 83] | 73 [61 to 83] | 76 [68 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 10 | 26
  Male | 24 | 29 | 53
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 40 | 39 | 79
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Netherlands | 40 | 39 | 79
NTproBNP [Median (Inter-Quartile Range); unit: pg/mL] | 4406 [2873 to 6979] | 6168 [3180 to 10489] | 4918 [3062 to 9555]

OUTCOME MEASURES:

1. Primary Outcome: Dyspnea
Description: Change in Dyspnea on VAS analogue scale (AUC)
  VAS Score is a measure/scale where patients on a scale from 0 to 100 can assign their current dyspnea score. 0 means there can be no worse dyspnea, 100 means it cannot get any better (perfect).
  The change in Dyspnea VAS means higher score is better outcomes.
  Individual changes in VAS score are be visualized (virtually) as a curve where the X-axis shows study day baseline to day 4, and y-axis shows VAS score. Using this approach, area under the curves for each study day (trapezoids) can be calculated, and added together, resulting in an overall VAS AUC score (mmxh) and change in VAS can be caculated
Time Frame: From baseline to Day 4
Measure: Mean (Standard Deviation); unit: mmxh
Arm/Group | Empagliflozin | Placebo
Number analyzed (Participants) | 37 | 36
mmxh | 1264 (1211) | 1650 (1240)
Statistical Analysis 1: Comparison: Empagliflozin vs Placebo; Test type: Superiority; p = 0.18, t-test, 2 sided

2. Primary Outcome: Diuretic Response
Description: Weight change from baseline per 40 mg of Furosemide equivalent
Time Frame: Total weight change from baseline to Day 4
Measure: Mean (Standard Deviation); unit: kg/40 mg Furosemide equivalent at day 4
Arm/Group | Empagliflozin | Placebo
Number analyzed (Participants) | 36 | 37
kg/40 mg Furosemide equivalent at day 4 | -0.35 (0.44) | -0.12 (1.52)
Statistical Analysis 1: Comparison: Empagliflozin vs Placebo; Test type: Superiority; p = 0.37, t-test, 2 sided

3. Primary Outcome: Length of Stay
Description: Hospital stay of Index admission
Time Frame: within 60 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Empagliflozin | Placebo
Number analyzed (Participants) | 39 | 38
days | 8 [6 to 10] | 8 [6 to 9]
Statistical Analysis 1: Comparison: Empagliflozin vs Placebo; Test type: Superiority; p = 0.58, Wilcoxon (Mann-Whitney)

4. Primary Outcome: Plasma NTproBNP
Description: Change in NTproBNP
Time Frame: From baseline to Day 4
Measure: Mean (Standard Deviation); unit: % change in NTproBNP at day 4
Arm/Group | Empagliflozin | Placebo
Number analyzed (Participants) | 37 | 34
% change in NTproBNP at day 4 | -46 (32) | -42 (31)
Statistical Analysis 1: Comparison: Empagliflozin vs Placebo; Test type: Superiority; p = 0.63, t-test, 2 sided

5. Secondary Outcome: Death and/or Heart Failure Re-admission
Description: Death and/or heart failure re-admission at day 30
Time Frame: Day 30
Measure: Count of Participants; unit: Participants
Arm/Group | Empagliflozin | Placebo
Number analyzed (Participants) | 40 | 39
Participants | 3 | 6
Statistical Analysis 1: Comparison: Empagliflozin vs Placebo; Test type: Superiority; p = 0.31, Regression, Logistic

6. Secondary Outcome: Inhospital Worsening Heart Failure, All Cause Mortality or Heart Failure Readmission at Day 60
Description: Inhospital Worsening Heart Failure or All Cause mortality or Heart Failure Readmission at day 60
Time Frame: 60 days
Measure: Count of Participants; unit: Participants
Arm/Group | Empagliflozin | Placebo
Number analyzed (Participants) | 40 | 39
Participants | 4 | 13
Statistical Analysis 1: Comparison: Empagliflozin vs Placebo; Test type: Superiority; p = 0.014, Regression, Logistic

7. Secondary Outcome: All Cause Mortality
Description: All Cause Mortality at 60 days
Time Frame: 60 day
Measure: Count of Participants; unit: Participants
Arm/Group | Empagliflozin | Placebo
Number analyzed (Participants) | 40 | 39
Participants | 1 | 3

8. Other Pre Specified Outcome: Serious Adverse Events
Description: SAE including all cause mortality. Per request Clintrials.gov different from Protocol definition
Time Frame: 60 days
Measure: Count of Participants; unit: Participants
Arm/Group | Empagliflozin | Placebo
Number analyzed (Participants) | 40 | 39
Participants
  Cardiovascular | 4 | 8
  Respiratory/Pulmonary | 0 | 1
  Renal/Urinary | 2 | 0
  Psychiatric | 0 | 1
  Infectious | 1 | 0
  Other | 1 | 0
  All Cause Mortality | 1 | 3

ADVERSE EVENTS:
Time Frame: 60 days
Arm/Group | Empagliflozin | Placebo
All-Cause Mortality (participants affected / at risk) | 1/40 | 3/39
Serious Adverse Events (participants affected / at risk) | 8/40 | 10/39
Other Adverse Events (participants affected / at risk) | 29/40 | 31/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Empagliflozin (N=40) | Placebo (N=39)
Worsening Heart Failure (Cardiac disorders) | 3 (3) | 4 (4)
Worsening Renal Function (General disorders) | 1 (1) | 0 (0)
Acute Kidney Injury (General disorders) | 1 (1) | 0 (0)
Angioedema (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hypovolemic shock (Cardiac disorders) | 0 (0) | 1 (1)
Delirium (General disorders) | 0 (0) | 1 (1)
Heart Failure (Cardiac disorders) | 0 (0) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
S. Aureus Bacteremia (Infections and infestations) | 1 (1) | 0 (0)
Syncope (Cardiac disorders) | 1 (1) | 1 (1)
Respiratory Failure (General disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Empagliflozin (N=40) | Placebo (N=39)
Cardiovascular (Blood and lymphatic system disorders) | 9 (9) | 17 (17)
Respiratory (General disorders) | 3 (3) | 2 (2)
Gastrointestinal (Gastrointestinal disorders) | 6 (6) | 9 (9)
Renal/Urinary (General disorders) | 15 (15) | 13 (13)
Metabolic (Metabolism and nutrition disorders) | 9 (9) | 9 (9)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 13 (13) | 13 (13)
Other (General disorders) | 6 (6) | 7 (7)

LIMITATIONS AND CAVEATS:
* Limited number of patients
* Screened many more patients then were included
* no standardized protocol for inhospital treatment for HF

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2017-10-20): https://cdn.clinicaltrials.gov/large-docs/60/NCT03200860/Prot_000.pdf
  • Statistical Analysis Plan (2019-09-03): https://cdn.clinicaltrials.gov/large-docs/60/NCT03200860/SAP_001.pdf